CLINICAL TRIAL: NCT02447315
Title: A Phase 1 Study to Investigate the Effect of Oral Doses of Pilocarpine on Salivary Secretion and Static Pupillometry in Healthy Subjects
Brief Title: A Study to Investigate the Effect of Oral Doses of Pilocarpine on Salivary Secretion and Static Pupillometry in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: TRAN-CL-0004; 2014-004753-13 (EudraCT Number)
Record Dates: First submitted 2015-03-31; First posted 2015-05-18 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Subjects
Keywords: Pilocarpine
MeSH Terms: interventions — Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Treatment Sequence ABCDD (Experimental): Subjects receive a single dose out of 4 oral doses of study drug (pilocarpine or matching placebo) per day for 5 subsequent days in the sequence ABCDD. Treatment A: pilocarpine low dose, Treatment B: pilocarpine medium dose, Treatment C: pilocarpine high dose, Treatment D: Placebo
  Interventions: Drug: Pilocarpine; Drug: Placebo
- Treatment Sequence BDACC (Experimental): Subjects receive a single dose out of 4 oral doses of study drug (pilocarpine or matching placebo) per day for 5 subsequent days in the sequence BDACC. Treatment A: pilocarpine low dose, Treatment B: pilocarpine medium dose, Treatment C: pilocarpine high dose, Treatment D: Placebo
  Interventions: Drug: Pilocarpine; Drug: Placebo
- Treatment Sequence CADBB (Experimental): Subjects receive a single dose out of 4 oral doses of study drug (pilocarpine or matching placebo) per day for 5 subsequent days in the sequence CADBB. Treatment A: pilocarpine low dose, Treatment B: pilocarpine medium dose, Treatment C: pilocarpine high dose, Treatment D: Placebo
  Interventions: Drug: Pilocarpine; Drug: Placebo
- Treatment Sequence DCBAA (Experimental): Subjects receive a single dose out of 4 oral doses of study drug (pilocarpine or matching placebo) per day for 5 subsequent days in the sequence DCBAA. Treatment A: pilocarpine low dose, Treatment B: pilocarpine medium dose, Treatment C: pilocarpine high dose, Treatment D: Placebo
  Interventions: Drug: Pilocarpine; Drug: Placebo

INTERVENTIONS:
Drug: Pilocarpine — oral
  Other Names: Salagen
Drug: Placebo — oral

SUMMARY:
The purpose of this study is to evaluate the pharmacodynamic effect of oral doses of pilocarpine on salivary secretion in healthy male and female subjects. In addition, pharmacodynamic effect on static pupillometry will be evaluated as well as pharmacokinetics and safety and tolerability of oral doses of pilocarpine in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Subject has a body mass index range of 18.5 to 30.0 kg/m2, inclusive. The subject weighs at least 50 kg. [screening]
* Female subject must either:

  * Be of nonchildbearing potential:

    1. Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
    2. Documented surgically sterile.
  * Or, if of childbearing potential:

    1. Agree not to try to become pregnant during the clinical study and for 28 days after the final study drug administration,
    2. Must have a negative serum pregnancy test at day -1,
    3. And, if heterosexually active, agree to consistently use 2 forms of highly effective birth control (at least 1 of which must be a barrier method) starting at screening and throughout the clinical study period after the final study drug administration. Highly effective forms of birth control include: Consistent and correct usage of established oral contraception; Injected or implanted hormonal methods of contraception; Established intrauterine device or intrauterine system; Barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository.
* Female subject must agree not to breastfeed starting at screening and throughout the clinical study period, and for 28 days after the final study drug administration.
* Female subject must not donate ova starting at screening and throughout the clinical study period, and for 28 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the clinical study period, and for 90 days after last study drug administration.
* Subject agrees not to participate in another interventional study while participation in the present clinical study, defined as signing the informed consent form until completion of the last study visit.

Exclusion Criteria:

* Female subject who has been pregnant within 6 months prior to screening assessment or breastfeeding within 3 months prior to screening.
* Subject has a known or suspected hypersensitivity to pilocarpine or any components of the formulation used.
* Subject has clinically significant, uncontrolled cardiorenal disease, uncontrolled asthma, chronic obstructive pulmonary disease, cholelithiasis, urolithiasis, current or previous peptic ulcer disease and/or any other chronic disease at risk for cholinergic agonists.
* Subject has a condition of the eye which could be affected by the intake of pilocarpine (e.g., acute iritis).
* Subject has any of the liver chemistry tests (aspartate aminotransferase [AST], alanine aminotransferase [ALT], alkaline phosphatase [ALP], gamma glutamyl transferase, total bilirubin [TBL]) above 1.5 × the upper limit of normal (ULN). In such a case, the assessment may be repeated once, on day -1.
* Subject has any clinically significant history of allergic conditions (including drug allergies, asthma, eczema or anaphylactic reactions, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* Subject has any history or evidence of any clinically significant cardiovascular, gastrointestinal, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease or malignancy.
* Subject has/had febrile illness or symptomatic, viral, bacterial (including upper respiratory infection) or fungal (noncutaneous) infection within 1 week prior to admission to the clinical unit (day -1).
* Subject has any clinically significant abnormality of the physical examination, ECG and clinical study protocol-defined clinical laboratory tests at screening or day -1.
* Subject has a mean pulse < 50 or > 90 bpm; mean systolic BP > 140 mmHg; mean diastolic BP > 90 mmHg (vital signs measurements taken in triplicate after subject has been resting in supine position for 5 minutes; pulse will be measured automatically) on admission to the clinical unit (day -1). If the mean BP exceeds the limits above, 1 additional triplicate can be taken.
* Subject has a mean corrected QT interval using Fridericia's formula (QTcF) > 430 ms (for male subjects) and > 450 ms (for female subjects) at screening. If the mean QTcF exceeds the limits above, 1 additional triplicate ECG can be taken on day -1.
* Subject uses any prescribed or nonprescribed drugs (including Salagen tablets or pilocarpine-containing eye drops in the month prior to first study drug administration / vitamins, natural and herbal remedies [e.g., St. John's wort] in the 2 weeks prior to first study drug administration) except for occasional use of paracetamol (up to 2 g/day) and except for use of contraceptives or hormone replacement therapy.
* Subject has a history of smoking within 1 month prior to first study drug administration (day 1).
* Subject has a history of drinking > 21 units of alcohol/week for male subjects or > 14 units of alcohol/week for female subjects (1 unit = 10 g pure alcohol = 250 mL of beer [5%] or 35 mL of spirits [35%] or 100 mL of wine [12%]) within 3 months prior to admission to the clinical unit (day -1).
* Subject has consumed grapefruit or Seville oranges or grapefruit- / Seville orange-containing products within 72 hours prior to admission to the clinical unit (day -1).
* Subject uses any inducer of metabolism (e.g., barbiturates, rifampin) within 1 month prior to admission to the clinical unit (day -1).
* Subject uses any drugs of abuse within 3 months prior to admission to the clinical unit (day -1).
* Subject had significant blood loss, donated 1 unit (500 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to admission to the clinical unit (day -1).
* Subject has a positive serology test for hepatitis B surface antigen, hepatitis A virus antibodies (immunoglobulin M), hepatitis C virus antibodies, or antibodies to human immunodeficiency virus type 1 (HIV-1) and/or type 2 (HIV-2) at screening.
* Subject participated in any clinical study or has been treated with any investigational drugs within 28 days prior to screening.
* Subject is an employee of the Astellas Group or Contract Research Organization (CRO).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2015-05; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameter salivary secretion at specified time points | Days 1-5
  Measure (mg/min) salivary secretion at specific timepoints
Pharmacodynamics assessed by area under the effect-time curve (AUE), saliva (AUEsal) | Days 1-5
Pharmacodynamics assessed by maximal effect (Emax), saliva (Emax, sal) | Days 1-5
Pharmacodynamics assessed by time at which the maximum salivary flow occurs (tmax, sal) | Days 1-5

SECONDARY OUTCOMES:
Pharmacodynamic profile pupil diameter pupS, pupLM, pupHM, AUEpupS, AUEpupLM, AUEpupHM, Emax,pupS, Emax,pupLM, Emax,pupHM, tmax,pupS, tmax,pupLM, tmax,pupHM | Days 1-5
  Pupil diameter, scotopic lighting condition (pupS); Pupil diameter, low mesopic lighting condition (pupLM); Pupil diameter, high mesopic lighting condition (pupHM); Area under the effect curve pupil diameter, scotopic lighting condition (AUEpupS); Area under the effect curve pupil diameter, low mesopic lighting condition (AUEpupLM); Area under the effect curve pupil diameter, high mesopic lighting condition (AUEpupHM); Maximum pharmacodynamic effect pupil diameter, scotopic lighting condition (Emax,pupS); Maximum pharmacodynamic effect pupil diameter, low mesopic lighting condition (Emax,pupLM); Maximum pharmacodynamic effect pupil diameter, high mesopic lighting condition (Emax,pupHM), Time at maximum concentration pupil diameter, scotopic lighting condition (tmax,pupS); Time at maximum concentration pupil diameter, low mesopic lighting condition (tmax,pupLM), Time at maximum concentration pupil diameter, high mesopic lighting condition (tmax,pupHM)
Safety profile assessed by adverse events, vital signs, routine electrocardiograms (ECG) , and clinical laboratory tests | up to Day 14
  Vital signs include body temperature, blood pressure and pulse. Clinical laboratory test include hematology, biochemistry and urinalysis.
Pharmacokinetics profile of pilocarpine: maximum concentration (Cmax), time of maximum concentration (tmax) and area under the concentration-time curve from the time of dosing (time zero) to 6 hours (AUC6) | Days 1-5

CONTACTS AND LOCATIONS:
Overall Officials: Associate Medical Director, Study Director — Astellas Pharma Europe B.V.
Locations (1):
- PAREXEL Early Phase Clinical Unit, Harrow, United Kingdom